CLINICAL TRIAL: NCT07167602
Title: Active Versus Positional Release Therapy in Athletes With Hamstring Shortening
Brief Title: Effect of Active and Positional Release on Hamstring Flexibility in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/I/REB/25/09/0060
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Hamstring Shortening, Short Hamstring Syndrome
Keywords: hamstring shortening, short hamstring syndrome, athlete, physiotherapy, manual therapy, active release therapy, positional release therapy

STUDY DESIGN:
Intervention Model Description: This study used a parallel assignment design in which 74 athletes with hamstring shortening were randomized into two equal groups. Group A received Positional Release Therapy combined with conventional physiotherapy, while Group B received Active Release Therapy combined with the same physiotherapy protocol.
Who Masked: Outcomes Assessor
Masking Description: This was a single-blinded trial. The outcomes assessor was blinded to group allocation and not involved in treatment delivery. Randomization was performed using sealed opaque envelopes, and group assignments were concealed from the assessor throughout data collection to minimize bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positional Release Therapy plus Conventional Physiotherapy (Experimental): Participants in this group first received conventional physiotherapy consisting of hot pack application (10 minutes), transcutaneous electrical nerve stimulation (15 minutes), passive hamstring stretching, and ankle pumps. After conventional therapy, Positional Release Therapy (PRT) was administered for the medial and lateral hamstrings. PRT involved positioning the muscle in shortened positions of comfort and applying gentle pressure with specific limb movements to facilitate relaxation, reduce neuromuscular tension, and relieve discomfort. Each session lasted approximately 50 minutes (35 minutes conventional therapy + 15 minutes PRT) and was delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Positional Release Therapy; Other: Conventional Physiotherapy
- Active Release Therapy plus Conventional Physiotherapy (Active Comparator): Participants in this group also received conventional physiotherapy consisting of hot pack application (10 minutes), transcutaneous electrical nerve stimulation (15 minutes), passive hamstring stretching, and ankle pumps. Following conventional care, Active Release Therapy (ART) was administered. ART involved applying longitudinal tension to the hamstring muscles while guiding the limb through specific ranges of motion, combined with brief isometric contractions of the hamstrings and quadriceps. This technique aimed to release adhesions, restore soft tissue mobility, and improve flexibility. Each session lasted approximately 50 minutes (35 minutes conventional therapy + 15 minutes ART) and was delivered twice weekly for 4 weeks.
  Interventions: Behavioral: Active Release Therapy; Other: Conventional Physiotherapy

INTERVENTIONS:
Behavioral: Positional Release Therapy — A manual therapy technique applied to the medial and lateral hamstrings after conventional physiotherapy. In PRT, the affected muscle is placed in a position of maximal comfort and relative shortening, while gentle pressure and controlled joint movements are applied. This position is held for approximately 30 seconds and repeated three times per session. The method aims to decrease neuromuscular tension, reduce pain, and promote muscle relaxation through a reflexive response. Distinct from Active Release Therapy, PRT does not involve active contractions or longitudinal tension but instead relies on positioning and relaxation to achieve therapeutic effects.
  Other Names: PRT; positional release technique
  Arms: Positional Release Therapy plus Conventional Physiotherapy
Behavioral: Active Release Therapy — A manual therapy technique applied to the hamstrings after conventional physiotherapy. ART combines therapist-applied longitudinal tension with patient movement and brief isometric contractions of both hamstrings and quadriceps. The limb is guided through specific ranges of motion to break down adhesions, restore tissue mobility, and improve flexibility. Unlike Positional Release Therapy, ART is an active technique requiring patient engagement through contractions and controlled movement against resistance, targeting scar tissue and myofascial restrictions.
  Other Names: ART; active release technique
  Arms: Active Release Therapy plus Conventional Physiotherapy
Other: Conventional Physiotherapy — Hot pack, TENS, hamstring stretching, ankle pumps (common to both groups).

SUMMARY:
Hamstring shortening is common in athletes and often causes pain, limited flexibility, and reduced function, which negatively impact performance. Manual therapy techniques such as Active Release Therapy (ART) and Positional Release Therapy (PRT) are frequently used, but their comparative effectiveness remains unclear.

This randomized, single-blinded clinical trial enrolled 74 athletes aged 18-35 years with hamstring shortening at the University of Lahore. Participants were randomly assigned to receive either PRT with conventional physiotherapy (hot pack, TENS, stretching, ankle pumps) or ART with the same physiotherapy protocol. Each group received two supervised sessions per week for four weeks.

The primary outcomes were pain (Numeric Pain Rating Scale), range of motion (Popliteal Angle), and functional ability (Lower Extremity Functional Scale). The Active Knee Extension test was used as a secondary outcome.

This study seeks to determine which manual therapy approach provides greater improvements in pain, flexibility, and function, with the goal of guiding evidence-based rehabilitation for athletes.

DETAILED DESCRIPTION:
Hamstring shortening, also referred to as short hamstring syndrome, is a frequent condition in athletes and has been linked to pain, reduced range of motion, and functional limitations that affect both sports performance and quality of life. Studies suggest that up to two-thirds of athletes may experience hamstring tightness, often as a result of repetitive strain, muscle imbalance, or inadequate recovery. Addressing this condition is therefore a priority in sports rehabilitation to minimize risk of injury and optimize performance.

Manual therapy is widely used in clinical practice to manage hamstring-related impairments. Among the commonly applied methods, Active Release Therapy (ART) aims to release adhesions and improve soft tissue mobility through tension and guided movements, while Positional Release Therapy (PRT) works by placing the muscle in a position of comfort to promote relaxation and reduce neuromuscular tension. Although both techniques have shown promise individually, limited evidence exists directly comparing their effectiveness in athletes with hamstring shortening.

This single-site, single-blinded randomized controlled trial was conducted at the University of Lahore Teaching Hospital to address this gap. Seventy-four athletes between 18 and 35 years of age were recruited using convenience sampling and randomized to one of two groups. Group A received Positional Release Therapy in addition to conventional physiotherapy, while Group B received Active Release Therapy with the same physiotherapy protocol. Conventional care included hot pack application, transcutaneous electrical nerve stimulation, hamstring stretching, and ankle pumps. Both groups received two sessions per week for four weeks, with outcome measures collected at baseline and post-intervention. The primary outcome measures were pain intensity, hamstring flexibility, and lower limb function, assessed respectively using the Numeric Pain Rating Scale (NPRS), Popliteal Angle test, and Lower Extremity Functional Scale (LEFS). The Active Knee Extension (AKE) test was included as a secondary outcome. The study design incorporated allocation concealment with sealed envelopes, blinding of assessors, and standardized protocols to minimize bias.

By directly comparing PRT and ART, this trial aims to provide evidence to guide clinical decision-making for the management of hamstring shortening in athletes. The results may inform physiotherapists, sports medicine professionals, and rehabilitation specialists about the relative benefits of each technique and support the use of effective, evidence-based interventions to improve pain, flexibility, and function in athletic populations.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age between 18 to 35
* Both genders
* Athletes with BMI between 18.5 kg/m² and 29.9 kg/m².
* Basketball, Football And Badminton Players.
* Athletes who practices atleast 3 days per week.
* Participants with Numeric pain rating scale values > 4.
* Participants with unilateral tightness of hamstring muscle with SLR < 80° and AKE < 125°

Exclusion Criteria:

* Participants with any acute chronic hamstring strain or lower back pain.
* Participants with leg length discrepancy.
* Participants with a sedentary lifestyle.
* Participants with upper motor neuron or lower motor neuron lesion.
* Participants with any previous history of lower extremity injury in the past three months
* Participants who are not willing to sign the consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Hamstring flexibility (Popliteal Angle test) | Baseline and 4 weeks after intervention
  Hamstring flexibility was assessed with a universal goniometer during the Popliteal Angle test. Participants lay supine with the hip flexed to 90°, and the knee was extended until a stretch was felt. The angle between the thigh and lower leg was recorded; larger angles reflect greater hamstring tightness. This test is widely used to quantify hamstring shortening.
Pain intensity (Numeric Pain Rating Scale, NPRS) | Baseline and 4 weeks (end of intervention)
  Pain severity in the posterior thigh was measured using the Numeric Pain Rating Scale (NPRS), an 11-point scale ranging from 0 ("no pain") to 10 ("worst imaginable pain"). Participants reported their average pain over the preceding 24 hours. This outcome captures the degree of symptom relief experienced after either Positional Release Therapy or Active Release Therapy.
Lower extremity function (Lower Extremity Functional Scale, LEFS) | Baseline and 4 weeks after intervention
  Functional ability was measured using the LEFS, a 20-item patient-reported questionnaire assessing difficulty with daily and sports-related lower limb activities. Each item is scored from 0 ("extreme difficulty or unable to perform") to 4 ("no difficulty"), for a total score range of 0-80. Higher scores indicate better function. The LEFS has high reliability (0.85-0.99) and validity for musculoskeletal conditions.

SECONDARY OUTCOMES:
Hamstring tightness (Active Knee Extension test, AKE) | Baseline and 4 weeks after intervention
  Hamstring tightness was measured with the Active Knee Extension (AKE) test using a universal goniometer. Participants lay supine with the hip flexed to 90° and the knee initially flexed to 90°. They were instructed to actively extend the knee until a stretch or mild pain was felt, and the angle was recorded. An angle >20° was classified as hamstring tightness. This test provides an active, participant-driven measure of flexibility, complementing the passive Popliteal Angle test.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asim Arif, Principal Investigator — University Institute of Physical Therapy, University of Lahore
Locations (1):
- University of Lahore - Teaching Hospital, University Institute of Physical Therapy, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
Can only be requested from principal investigator